CLINICAL TRIAL: NCT03985098
Title: A Motivational Interviewing Intervention Customized by Patient Adherence Patterns
Brief Title: Motivational Interviewing (MI) Intervention to Improve Adherence
Acronym: MI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Susan Abughosh,, Associate Professor, University of Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00000718; R15HL135700-01A1 (NIH)
Record Dates: First submitted 2019-06-10; First posted 2019-06-13 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
Keywords: Motivational interviewing; trajectory modeling; medication adherence
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motivational interviewing intervention arm (Experimental): The intervention will be a phone call by a pharmacy student that will use MI strategies to identify and address the adherence barrier(s) and 5 monthly follow up calls
  Interventions: Behavioral: Motivational interviewing intervention arm
- Control (No Intervention): usual care

INTERVENTIONS:
Behavioral: Motivational interviewing intervention arm — The intervention will be a phone call by a pharmacy student that will use MI strategies to identify and address the adherence barrier(s) and 5 monthly follow up calls
  Arms: Motivational interviewing intervention arm

SUMMARY:
The purpose of this study is to examine the effectiveness of a telephone motivational interviewing intervention by pharmacy students in enhancing adherence to angiotensin converting enzyme inhibitors (ACEI)/ angiotensin receptor blockers (ARB) (ACE/ARBs) among patients with diabetes and hypertension in a Medicare advantage plan.

DETAILED DESCRIPTION:
Angiotensin converting enzyme inhibitors (ACEI)/ angiotensin receptor blockers (ARB) are highly recommended for patients with both diabetes (DM) and hypertension (HTN), and their efficacy in reducing macrovascular and microvascular complications of DM is well-documented. Poor adherence remains a significant barrier to achieving full effectiveness and optimal long-term outcomes. This study aims to develop innovative group-based trajectory models to identify patients with similar ACE/ARB medication filling behavior among patients with co-morbid HTN and DM. The proportion of days covered (PDC), often used as an adherence measure, reduces complex patterns of longitudinal observations into a single value that cannot adequately depict different adherence experiences. Group based trajectory models are designed to identify patients with similar longitudinal patterns while capturing the dynamic nature. A motivational interviewing (MI) pharmacy student telephone intervention will then be customized by the identified trajectories and tested to demonstrate effectiveness in enhancing adherence. In pilot work, the investigator's team has demonstrated improvements in adherence through a pharmacy student telephone MI intervention. Pharmacy students have the knowledge base and training to provide comparable services to pharmacists at a lower cost. MI fosters behavior change by setting desired goals and promoting self-efficacy in a supportive, collaborative way. The objectives are to 1. Develop group-based trajectory models to identify patients with similar medication filling behavior patterns among patients enrolled in a Medicare advantage plan and 2. Customize an MI pharmacy student telephone intervention by the adherence patterns identified, and demonstrate the benefit of the customized intervention in improving adherence. Phase 1 of the project will be a retrospective analysis of 12 month refill data to determine patient adherence patterns. Phase 2 will be a prospective study among non-adherent patients to evaluate the effectiveness of the customized intervention (n=500). The students will contact patients assigned to the intervention group and follow a protocol using the Ask-Provide-Ask approach of MI given the patient adherence pattern for a tailored education. Monthly follow-up calls will be carried out for 6 months. Adherence during the 6 and 12 months post-intervention will be evaluated for the intervention and control groups as PDC as well as a categorical variable. Chi-square and t-tests will be used to evaluate the intervention effect. Multivariable multiple and logistic regression will be carried out in case of any significant differences in baseline characteristics. Implementing this project will provide students a unique MI training as a new way of communicating with patients. The training is further strengthened by PhD students trained in research design and statistical analyses to assist in the automated data analysis. The project will formulate a strong adherence research team at University of Houston that will be instrumental in implementing customized innovative interventions to improve medication adherence and subsequent health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Continuous enrollment over the study period July 2016 to December 2018.
2. A prescription filled for an ACEI or ARB medication between July 1st, 2017- December 31st, 2017. This will be defined as the index date (for phase 1).
3. Diagnosis of both DM and HTN prior to index date, identified through the health plan's medical claims program (CCMS) using the International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) codes only.

Exclusion Criteria:

1. Disenrollment from drug plan.
2. Death prior to end of the study.
3. Having a diagnosis of dementia in the one-year pre-index period.
4. Having an ACEI/ARB contraindication like angioedema, hyperkalemia, and renal artery stenosis in the one-year pre-index period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 727 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2022-03-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Omar Serna, Houston, Texas, United States

REFERENCES:
- [Derived] Mohan A, Majd Z, Johnson ML, Essien EJ, Barner J, Serna O, Gallardo E, Fleming ML, Ordonez N, Holstad MM, Abughosh SM. A Motivational Interviewing Intervention to Improve Adherence to ACEIs/ARBs among Nonadherent Older Adults with Comorbid Hypertension and Diabetes. Drugs Aging. 2023 Apr;40(4):377-390. doi: 10.1007/s40266-023-01008-6. Epub 2023 Feb 27. PMID 36847995

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Motivational Interviewing Intervention Arm | Control
Started | 247 | 480
Completed | 240 | 480
Not Completed | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing Intervention Arm | Control | Total
Number analyzed (Participants) | 240 | 480 | 720
Age, Customized [Count of Participants; unit: Participants]
  Age: <70 years | 123 | 257 | 380
  Age: ≥70 years | 117 | 223 | 340
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 272 | 417
  Male | 95 | 208 | 303
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 240 | 480 | 720
health plan [Count of Participants; unit: Participants]
  Low-income subsidy | 118 | 236 | 354
  No-subsidy | 122 | 244 | 366
prescriber specialty [Count of Participants; unit: Participants]
  General | 207 | 410 | 617
  Specialty | 27 | 54 | 81
  Missing | 6 | 16 | 22
refill type [Count of Participants; unit: Participants]
  <90 days | 26 | 55 | 81
  ≥90 days | 214 | 425 | 639
Comorbidities [Count of Participants; unit: Participants]
  Myocardial infarction: Yes | 4 | 10 | 14
  Myocardial infarction: No | 236 | 470 | 706
  Depression: Yes | 31 | 56 | 87
  Depression: No | 209 | 424 | 633
  Congestive heart failure: Yes | 26 | 30 | 56
  Congestive heart failure: No | 214 | 450 | 664
  Stroke: Yes | 10 | 18 | 28
  Stroke: No | 230 | 462 | 692
  Coronary artery disease: Yes | 63 | 92 | 155
  Coronary artery disease: No | 177 | 388 | 565
number of concomitant medications [Count of Participants; unit: Participants]
  ≤2 | 169 | 340 | 509
  >2 | 71 | 140 | 211
regimen complexity [Mean (Standard Deviation); unit: scores on a scale] — Regimen complexity was defined as number of prescribed doses per day multiplied by number of medications as determined on index date. It is a continuous variable that could take any value. (observed range: 0.5-47) Existing literature has been inconsistent with the association between regimen complexity and adherence (negative and positive associations). Therefore, we decided to control for it in the model, however, we did not find any significant association (p=0.54). In other words, every unit increase in "regimen complexity" did not have an impact on the study outcome.
  scores on a scale | 4.27 (4.32) | 3.86 (3.94) | 3.99 (4.07)
prevalent users [Count of Participants; unit: Participants] — Prevalent users were defined as patients who were prescribed ACEI/ARB medications during the 6-months baseline period.
  Participants
    No | 25 | 90 | 115
    Yes | 215 | 390 | 605
prior hospitalizations [Count of Participants; unit: Participants]
  ≥1 | 26 | 45 | 71
  None | 214 | 435 | 649
CMS risk score [Mean (Standard Deviation); unit: scores on a scale] — The CMS risk score accounts for disease severity and medication burden. It is comprised of 189 disease classifications used in risk adjustment of clinical outcomes in Medicare populations. This variable could take any value within a continuous range. (observed range: 0.25-6.00) The existing literature presents conflicting evidence on the relationship between adherence and risk score (positive or negative). However, we did not find any significant association (p=0.33). In other words, every unit increase in "CMS risk score" did not have an impact on the study outcome.
  scores on a scale | 1.50 (0.99) | 1.36 (0.83) | 1.41 (0.89)

OUTCOME MEASURES:

1. Primary Outcome: Adherence Measure
Description: Proportion of days covered (PDC): measured by examining refill data, both as a continuous measure as well as a categorical measure with a PDC of 0.8 or more considered adherent. It ranges from 0-1.
Time Frame: 12 months following initial call
Measure: Mean (Standard Error); unit: Proportion of days covered
Arm/Group | Motivational Interviewing Intervention Arm | Control
Number analyzed (Participants) | 240 | 480
Proportion of days covered | 0.63 (0.34) | 0.56 (0.35)

ADVERSE EVENTS:
Time Frame: Up to 12 months from initial call
Description: This study does not involve more than Minimal Risk for the safety of patients. The intervention involves only a phone call to educate the patient about adherence and participation is completely based on the patient's consent. They can withdraw or choose to stop the call at any point. Thus, it is not anticipated that the intervention can harm any patient in any way.
Arm/Group | Motivational Interviewing Intervention Arm | Control
All-Cause Mortality (participants affected / at risk) | 0/240 | 0/480
Serious Adverse Events (participants affected / at risk) | 0/240 | 0/480
Other Adverse Events (participants affected / at risk) | 0/240 | 0/480

LIMITATIONS AND CAVEATS:
While the initial plan for the intervention was to have monthly follow-up calls, due to the COVID-19 pandemic, there were gaps in the intervention, which could have affected the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT03985098/Prot_SAP_000.pdf